CLINICAL TRIAL: NCT06857500
Title: Brentuximab Vedotin with Adriamycin, Vinblastine and Dacarbazine for Patients Aged 18-59 Years with Untreated Advanced-stage Classical Hodgkin Lymphoma: a Real-life Experience
Acronym: FED_RealBV
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Marco Picardi, Full Professor, Federico II University
Other Study IDs: FED_RealBV
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Classic Hodgkin Lymphoma; Advanced Hodgkin Lymphoma
Keywords: classic Hodgkin Limphoma; advanced stages; 18-59

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Classical Hodgkin lymphoma (cHL) is commonly diagnosed in young adults and adults (YP&A) defined by the National Cancer Institute as 18 to 59 years of age. Clinically, these patients often present with poor prognostic factors such as advanced stage. In phase III trials that primarily include patients aged 18 to 59 years, several international cooperative oncology groups have studied new initial treatments for Ann Arbor stage III and IV cHL. These treatments include traditional dose-dense/dose-intensity cytotoxic approaches (such as the FONDAZIONE ITALIANA LINFOMI FIL-ROUGE trial) or novel selectively active agents such as nivolumab (SWOG S1826 trial) or brentuximab vedotin (BV) (HD21 and ECHELON-1 trials). Among these, the most beneficial initial treatment schedule remains controversial, not only because of additional acute toxicities and additional drug-related expenses, but especially for long-term disease control.

Brentuximab Vedotin is a monoclonal antibody conjugated with a protease-cleavable linker to the microtubule disrupting agent monomethylauristatin E, which targets CD30 on Reed-Sternberg cells. The global phase III ECHELON-1 study compared BV in combination with adriamycin, vinblastine, and dacarbazine (BV+AVD) versus adriamycin, bleomycin, vinblastine, and dacarbazine (ABVD) in patients with newly diagnosed stage III and IV cHL.

Among the 1,334 patients included, the majority of cases (1,148; 86%) were YP&A age. At the 51st National Congress of the Italian Society of Hematology, a post-hoc analysis of long-term follow-up data from ECHELON-1 was conducted to assess progression-free survival (PFS) in the subgroup aged 18 to 59 years. YP&A patients received either BV+AVD (N= 580) or ABVD (N= 568): after 2 years of follow-up, the Kaplan-Mayer curve of PFS for BV+AVD flattened with a plateau that remained consistently at 87% up to 7 years with a number of events of 67 compared to the Kaplan-Mayer curve of PFS for ABVD that decreased during follow-up to 79% with a number of 91 events (HR 0.667; 95% CI: 0.486-0.914; P= 0.011 by log-rank test). Based on the study design, no patients in either arm received consolidation radiotherapy to residual nodal masses (RNM). Low rates of second malignancies (5% for BV+AVD vs. 6% for ABVD), no apparent effect on fertility (pregnancies: 92 for BV+AVD vs. 73 for ABVD), and resolution or improvement of peripheral neuropathy in the majority of patients were reported by the investigators. Additionally, the YP&A subgroup showed a 7-year overall survival of 97% (number of events, 21) for BV+AVD vs. 92% (number of events, 39) for ABVD (HR, 0.489; 95% CI, 0.287-0.833; P= 0.007 by log-rank test) with a 51% reduction in the risk of death from any cause 13 . These data underscore the clinical benefit of BV+AVD for patients aged 18-59 years, mainly regarding disease cure, with no new safety signals. Therefore, BV+AVD is one of the standards of care for YP&A with untreated advanced cHL.

To date, there have been no studies outside of prospective clinical trials examining the efficacy and safety of BV+AVD for newly diagnosed advanced cHL in patients aged 18-59 years. In this study, involving 3 Italian oncology centers dedicated to the care of HL, we aim to examine a cohort of YP&A with stage III-IV cHL with a median follow-up of two years after first-line treatment with BV+AVD, with the aim of understanding the outcome and specific side effects in a real-life experience.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of previously untreated c-HL
* stage III or IV at diagnosis
* treatment with at least one cycle of therapy according to the Brentuximab Vedotin + AVD regimen
* age between 18 and 59 years
* ECOG at diagnosis: PS 0-3
* negative HIV test
* follow up from the end of treatment >24 months All diagnoses are made according to the WHO classification of Lymphomas.

Exclusion Criteria:

* Creatinine clearance <30 ml/min at diagnosis
* transaminase >3 ULN at diagnosis
* absolute neutrophil count >500/mmc at diagnosis
* hemoglobin concentrations <9 g/dL at diagnosis
* platelet count <75000/mmc at diagnosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 19-60 year old c-HL patients, previously untreated with Ann Arbor stage III or IV. ECOG PS 0-3, GLS ≥-20% at echocardiographic assessment and human immunodeficiency virus negativity.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | from 1 January 2013 to 1 January 2025
  The primary endpoint was the activity of the Brentuximab Vedotin- based front-line strategy in terms of OS.

SECONDARY OUTCOMES:
Progression-free survival | from 1 January 2013 to 1 January 2025
  Progression free survival
adverse events | from 1 January 2013 to 1 January 2025
  grade >3 adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University,, Naples, Italy, Italy

REFERENCES:
- [Derived] Picardi M, Vincenzi A, Giordano C, Pugliese N, Scarpa A, Lombardi A, Vigliar E, Troncone G, Cappiello R, Mascolo M, Esposito G, Prastaro M, Santoro C, Esposito R, Tocchetti CG, Mainolfi C, Fonti R, Del Vecchio S, Trastulli F, Annunziata M, Iula R, Califano C, Carchia M, Persico M, Salemme A, Nicolai E, Soricelli A, Salvatore M, Pane F. Brentuximab Vedotin With Adriamycin, Vinblastine, and Dacarbazine for Patients Aged 18-59 Years With Untreated Advanced Stage Classical Hodgkin Lymphoma: The Largest Real-Life Series From Southern Italy Cancer Centers. Eur J Haematol. 2026 Feb;116(2):174-184. doi: 10.1111/ejh.70060. Epub 2025 Nov 6. PMID 41198414